CLINICAL TRIAL: NCT01929200
Title: Randomized, Open-label, Multicenter Study of Icotinib as Adjuvant Therapy in Treating Stage II-IIIA Non-small-cell Lung Cancer Patients With Positive EGFR Mutation
Brief Title: Icotinib as Adjuvant Therapy in Treating Non-small-cell Lung Cancer Patients With Positive EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV50
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Therapeutics; icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-year treatment with icotinib (Experimental): Patients will receive 1-year treatment with icotinib after operation.
  Interventions: Drug: 1-year treatment with icotinib
- 2-year treatment with icotinib (Experimental): Patients will receive 2-year treatment with icotinib after operation.
  Interventions: Drug: 2-year treatment with icotinib

INTERVENTIONS:
Drug: 1-year treatment with icotinib — Icotinib is administered orally with a dose 125 mg 3 times daily within 4-6 weeks after operation for 1 year.
  Other Names: Commana; BPI-2009
  Arms: 1-year treatment with icotinib
Drug: 2-year treatment with icotinib — Icotinib is administered orally with a dose 125 mg 3 times daily within 4-6 weeks after operation for 2 years.
  Other Names: Commana; BPI-2009
  Arms: 2-year treatment with icotinib

SUMMARY:
This study is designed to evaluate the efficacy of icotinib as adjuvant therapy in treating such patients. The primary endpoint is to compare the recurrence-free survival after 1-year or 2-year treatment with icotinib.

DETAILED DESCRIPTION:
Adjuvant therapy has been proved effective in treating stage II-IIIA non-small-cell lung cancer. However, few data on the treating time of adjuvant therapy is available. Here we conduct a randomized, prospective study to compare the recurrence-free survival after 1-year or 2-year treatment with icotinib in EGFR-mutated non-small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the written informed consent
* The patients present with operable stage II-IIIA non-small-cell lung cancers with 19 or 21 exon mutation
* The patients have no history of anti-cancer therapies including chemotherapy, radiation therapy
* The patients' Eastern Cooperative Oncology Group scores are ≤ 0-2

Exclusion Criteria:

* Patients with unresected tumor
* Wild EGFR type
* Allergic to the study drug
* Patients have severe non-cancerous diseases
* Patients are undergoing current administration of anti-cancer therapies, or are attending some other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival | 6 months

SECONDARY OUTCOMES:
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yue Yang, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer hospital, Beijing, China

REFERENCES:
- [Background] Lv C, Ma Y, Feng Q, Fang F, Bai H, Zhao B, Yan S, Wu N, Zheng Q, Li S, Chen J, Wang J, Feng Y, Wang Y, Pei Y, Fang J, Yang Y. A pilot study: sequential gemcitabine/cisplatin and icotinib as induction therapy for stage IIB to IIIA non-small-cell lung adenocarcinoma. World J Surg Oncol. 2013 Apr 26;11:96. doi: 10.1186/1477-7819-11-96. PMID 23621919
- [Derived] Lv C, Wang R, Li S, Yan S, Wang Y, Chen J, Wang L, Liu Y, Guo Z, Wang J, Pei Y, Yu L, Wu N, Lu F, Gao F, Chen J, Liu Y, Wang X, Li S, Han B, Zhang L, Ma Y, Ding L, Wang Y, Yuan X, Yang Y. Randomized phase II adjuvant trial to compare two treatment durations of icotinib (2 years versus 1 year) for stage II-IIIA EGFR-positive lung adenocarcinoma patients (ICOMPARE study). ESMO Open. 2023 Aug;8(4):101565. doi: 10.1016/j.esmoop.2023.101565. Epub 2023 Jun 20. PMID 37348348